CLINICAL TRIAL: NCT06008639
Title: Efficacy and Safety of Near Infrared Light Therapy for Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Danyang Huichuang Medical Equipment Co., Ltd. (Industry)
Collaborators: Rehabilitation Hospital Affiliated to National Research Center for Rehabilitation Technical Aids (Unknown); First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018YFC2001700
Record Dates: First submitted 2023-06-15; First posted 2023-08-23 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Mild to Moderate Alzheimer's Disease

STUDY DESIGN:
Intervention Model Description: The subjects will be randomly assigned to the treatment group or the control group for 30 minutes/day (5-6 days a week) for 4 months while the treatment group is active settings and the control group is sham settings.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Active Comparator): active setting
  Interventions: Device: treatment group-Device: NirsCure - Active NirsCure - Active settings
- Control group (Placebo Comparator): sham setting
  Interventions: Device: placebo group-Device: NirsCure - Sham NirsCure - Sham settings

INTERVENTIONS:
Device: treatment group-Device: NirsCure - Active NirsCure - Active settings — Treatment was performed once a day,5-6 times a week for 16 weeks.
  Arms: treatment group
Device: placebo group-Device: NirsCure - Sham NirsCure - Sham settings — Treatment was performed once a day,5-6 times a week for 16 weeks.
  Arms: Control group

SUMMARY:
To explore the efficacy and safety of near infrared light therapy for Alzheimer's disease. Each subject will be numbered and their medical records will be established. The subjects will be randomly assigned to the treatment group or the control group for 30 minutes/day (5-6 days a week) for 4 months while the treatment group is active settings and the control group is sham settings.Follow-up visits will be conducted at 2 months, 4 months and 2 months after treatment. At each follow-up, scale assessment, blood, MRI, and EEG were observed

ELIGIBILITY:
Inclusion Criteria:

* The age of registration is 50-85 years old, male or female.
* The MMSE score < 26 points can be used to complete the scale assessment.
* Patients who are not on medication and who are taking psychotropic or cognitive-improving drugs must have a stable dose for at least 12 weeks before the trial and remain the same for the duration of treatment.
* Agree to participate in the clinical trial, willing to maintain the original treatment plan during the trial, and have signed the informed consent

Exclusion Criteria:

* MRI showed evidence of abnormalities other than Alzheimer's disease, such as cerebral infarction at key sites and severe leukodystrophy (Fezakas>Level 3).
* There are contraindications to MRI scanning, such as metal implants, claustrophobia, etc.
* A history of stroke or seizures.
* Photosensitive to sunlight or visible light, eczema or increased sensitivity of the skin at the treatment site.
* Severe vision or hearing impairment.
* Alcohol dependence, drug or other drug addiction or addiction tendency.
* During the study , subjects were pregnant, breastfeeding, or planning to pregnancy.
* He/She is currently participating in another study related to the treatment of AD.
* Researchers think that participants could not be included.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ADAS-cog | 8 weeks, 16 weeks and 24 weeks
  Alzheimer's Disease Assessment Scale - Cognitive section ,ADAS-Cog；The higher the score, the worse.
Change from baseline in MMSE | 8 weeks, 16 weeks and 24 weeks
  (Mini-Mental State Examination, MMSE ;The higher the score, the better.
Change from baseline in ALFF | 8 weeks, 16 weeks and 24 weeks
  The amplitudeof low-frequency fluctuations, ALFF;The increase of ALFF indicates that neuronal excitability and metabolism are enhanced, while the decrease of ALFF indicates that neuronal spontaneous activity is inhibited.

SECONDARY OUTCOMES:
Change from baseline in MOCA | 8 weeks, 16 weeks and 24 weeks
  Montreal Cognitive Assessment, MoCA；The higher the score, the better.
Change from baseline in ADCS-CGIC | 8 weeks, 16 weeks and 24 weeks
  Alzheimer's Disease Cooperative study-clinical global impression of change scale，ADCS-CGIC
Change from baseline in ADCS-ADL | 8 weeks, 16 weeks and 24 weeks
  Alzheimer's Disease Cooperative study-Activities of Daily Living Scale，ADCS-ADL;The higher the score, the better.
Change from baseline in NPI | 8 weeks, 16 weeks and 24 weeks
  Neuropaychiatic Inventory，NPI；The higher the score, the worse.
Change from baseline in HAMD | 8 weeks, 16 weeks and 24 weeks
  Hamilton depression scale,HAMD; The higher the score, the worse.
Aβ amyloid and tau levels | 8 weeks, 16 weeks and 24 weeks
  Plasma Aβ and Tau proteins are thought to be related to the pathogenesis of AD; The lower the protein level, the better.
MRI | 8 weeks, 16 weeks and 24 weeks
  Magnet Resonance Imaging,MRI; The brain volume, hippocampus volume, links between brain regions will be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Ze Lv, Principal Investigator — Rehabilitation Hospital Affiliated to National Research Center for Rehabilitation Technical Aids
Locations (2):
- China (2):
  - Rehabilitation hospital affiliated National Research Center for Rehabilitation Technical Aids, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Sichuan

IPD SHARING:
Plan to Share IPD: No